CLINICAL TRIAL: NCT05355077
Title: An Open-label, Dose-Escalation, Multiple-Dose Phase 1 Clinical Study to Evaluate the Pharmacokinetics, Safety and Tolerability of JT001 Tablets in Caucasian Healthy Subjects After Oral Administrations
Brief Title: Evaluate the Pharmacokinetics, Safety and Tolerability of JT001 Tablets
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Development strategy adjustment
Sponsor: Shanghai Vinnerna Biosciences Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: JT001-005-I
Record Dates: First submitted 2022-04-20; First posted 2022-05-02 (Actual); Last update posted 2023-02-09 (Actual); Status verified 2022-04

CONDITIONS: Healthy Subjects
MeSH Terms: interventions — GS-621763; BID protein, human

STUDY DESIGN:
Intervention Model Description: Sequential
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group 1 (Experimental): JT001 (VV116):200 mg, oral, Twice a day
  Interventions: Drug: JT001 200mg Bid
- Group 2 (Experimental): JT001 (VV116):400 mg, oral, Twice a day
  Interventions: Drug: JT001 400mg Bid
- Group 3 (Experimental): JT001 (VV116):600 mg, oral, Twice a day
  Interventions: Drug: JT001 600mg Bid

INTERVENTIONS:
Drug: JT001 200mg Bid — JT001 (VV116):200 mg,oral,Twice a day,6 consecutive days and the last administration will be given in the morning on Day 6
  Other Names: VV116
  Arms: Group 1
Drug: JT001 400mg Bid — JT001 (VV116):400 mg,oral,Twice a day,6 consecutive days and the last administration will be given in the morning on Day 6
  Other Names: VV116
  Arms: Group 2
Drug: JT001 600mg Bid — JT001 (VV116):600 mg,oral,Twice a day,6 consecutive days and the last administration will be given in the morning on Day 6
  Other Names: VV116
  Arms: Group 3

SUMMARY:
This is a Phase 1, open-label, dose-escalation, multiple-dose study to investigate pharmacokinetics and safety of JT001 (VV116) in Caucasian healthy subjects.

DETAILED DESCRIPTION:
Subjects will be admitted to the Phase 1 clinical study ward on the day before administration (Day -1, baseline phase), and will be confined until all examinations and assessments are completed on Day 8. Subjects will be followed up on Day 12 (± 1 day); if there are abnormalities, an unscheduled visit may be arranged for subjects at the Investigators discretion. Subjects who withdraw early should be encouraged to complete the early withdrawal visit.

At the Screening visit, subjects who are willing to take part in the study will sign informed consent forms (ICFs) and complete the screening examinations. Subjects who meet all of the inclusion criteria and none of the exclusion criteria will be assigned to receive the investigational product (IP) at 1 of the 3 doses according to the dose-escalation scheme, and will be followed up until the 6th day after the last administration.

Time of Collection of PK Blood Samples

To gather the PK data, PK blood samples will be collected at the following specified times:

Day 1: pre-dose (within 1 h before the first administration), and at 10 min, 20 min, 30 min, 45 min, 1 hour, 1.5 hours, 2 hours, 3 hours, 4 hours, 6 hours, 8 hours, and 12 hours after the first administration.

Day 5: pre-dose (within 0.5 hour before each administration) Day 6: pre-dose (within 0.5 hour before administration), and at 10 min, 20 min, 30 min, 45 min, 1 hour, 1.5 hours, 2 hours, 3 hours, 4 hours, 6 hours, 8 hours, 12 hours, 24 hours, and 48 hours post-dose.

Dose-Escalation Scheme This study consists of 3 dosing group (200, 400, and 600 mg). A dose-escalation design is used, sequentially from the low-dose group to the high-dose group, and each subject will only receive oral administration at one dose level according to the dose-escalation scheme. All subjects will be administered orally twice a day (approximately 12 hours apart) for 6 consecutive days and the last administration will be given in the morning on Day 6. All doses must be taken under fasting conditions.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy Caucasian male or female (excluding Middle East) subjects aged 18 to 55 years (inclusive at the time of informed consent). Caucasians are defined as subjects who have 2 parents of Caucasian/European ancestry and 4 grandparents of Caucasian/European ancestry.
2. Subjects must have a Body Mass Index (BMI) ≥ 18.0 and ≤ 32.0 kg/m2 at Screening with body weight: male ≥ 50 kg, female ≥ 45 kg.
3. Subjects must be in good general health, have no clinically significant abnormalities on vital signs, physical examination, laboratory test, ophthalmology, and ECG at Screening and/or before administration of the initial dose of the study drug.
4. Women of childbearing potential (WOCBP) must have a negative serum or urine pregnancy test within 24 hours prior to the start of study drug and must not be breastfeeding, lactating or planning pregnancy during the study period. WOCBP are defined as any female who has experienced menarche and who has not undergone surgical sterilization (hysterectomy or bilateral oophorectomy) and is not postmenopausal. Menopause is defined as 12 months of amenorrhea in the absence of other biological causes. In addition, females under the age of 55 years must have a documented serum follicle stimulating hormone (FSH) level > 40mIU/mL to confirm menopause. Male participants with potentially postmenopausal partners who are under the age of 55 years must use condoms unless their partner's postmenopausal status has been confirmed by FSH level.
5. Subjects must be willing and able to provide written informed consent after the nature of the study has been explained and before the commencement of any study procedures.

Exclusion Criteria:

1. Known history of allergy to the study drug.
2. History of severe allergic or anaphylactic reactions.
3. Subjects with confirmed diseases in the central nervous system, cardiovascular system, digestive system, respiratory system, urinary system, blood system, metabolic disorders, etc., and require medical intervention, or other diseases that are not suitable for participating in clinical studies (such as psychiatric history, etc.). Subjects with mild depression and anxiety may be enrolled if stable and not medicated.
4. Medical history considered by the Investigator to impact the assessment of PK profiles.
5. Blood donation or blood loss ≥ 400 mL before screening or has used blood products. Subjects who have donated blood within 1 month or plasma donation within 7 days of Screening will not be included in the study.
6. Subjects who have received treatment with another investigational drug within 3 months of screening or is participating in another study at the time of screening.
7. Use of any prescription drugs, over the counter (OTC) medication, herbal remedies, supplements, or vitamins within 1 week before screening. Taking paracetamol (up to 2000 mg/day) is allowed.
8. Subjects with alcohol addiction within 1 year before screening, defined as drinking more than 14 units per week (1 unit is equivalent to approximately 200 mL of beer with 5% alcohol content, or 25 mL of spirits with 40% alcohol content, or 85 mL of wine with 12% alcohol content).
9. Subjects who have a history of smoking more than 10 cigarettes a day or the equivalent amount within 1 year before screening will not be included. Light smoking (e.g., 10 cigarettes/week) within 1 month prior to screening is acceptable as long as the participant is willing to abstain from smoking during inpatient stay.
10. Subject is unwilling to abstain from smoking or alcohol during the study.
11. Positive test for hepatitis B surface antigen (HBsAg), hepatitis C virus antibody (Anti-HCV), Treponema pallidum antibody, and human immunodeficiency virus (HIV) antibody at Screening.
12. Subjects with abnormal ALT or AST value that is considered clinically by the Investigator at Screening will not be included in the study.
13. Glomerular filtration rate (eGFR) < lower limit of normal (LLN) at Screening. The CKD-EPI formula will be used for the eGFR calculation.
14. Abnormal ECG findings considered by the Investigator to be clinically significant, single-examination QTcF (heart rate corrected) > 450 ms in males and > 470 ms in females, and/or other clinically significant abnormalities at Screening.
15. Pregnant or lactating at Screening or planning to become pregnant (self or partner) from Screening until 3 months after the last administration of the study drug.
16. Subject is considered to have other factors, in the opinion of the Investigator, which would make it unlikely that the subject will comply with the protocol or complete the study per protocol.
17. Subjects who received any COVID-19 vaccination within 14 days prior to the first administration of the study drug will not be included in the study.
18. Any other condition that would, in the Investigator's judgement, contraindicate the patient's participation in the clinical study due to safety concerns or compliance with clinical study procedures or interpretation of study results.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2022-05-02 (Estimated); Primary Completion 2022-08-01 (Estimated); Study Completion 2022-10-24 (Estimated)

PRIMARY OUTCOMES:
To explore the pharmacokinetics of JT001 and its prominent metabolite 116-N1 in Caucasian healthysubjects | Day 1,Day 5,Day 6:until 48 hours post-dose.
  Pharmacokinetic (PK) parameters: peak concentration (Cmax) of JT001 (VV116) and its metabolite 116-N1.
To explore the pharmacokinetics of JT001 and its prominent metabolite 116-N1 in Caucasian healthysubjects | Day 1,Day 5,Day 6:until 48 hours post-dose.
  Pharmacokinetic (PK) parameters : time to peak concentration (Tmax) of JT001 (VV116) and its metabolite 116-N1.
To explore the pharmacokinetics of JT001 and its prominent metabolite 116-N1 in Caucasian healthysubjects | Day 1,Day 5,Day 6:until 48 hours post-dose.
  Pharmacokinetic (PK) parameters: trough concentration (Ctrough) of JT001 (VV116) and its metabolite 116-N1.
To explore the pharmacokinetics of JT001 and its prominent metabolite 116-N1 in Caucasian healthysubjects | Day 1,Day 5,Day 6:until 48 hours post-dose.
  Pharmacokinetic (PK) parameters: area under the plasma concentration-time curves (AUC0-t, AUC0-∞, and AUC0-τ) of JT001 (VV116) and its metabolite 116-N1.
To explore the pharmacokinetics of JT001 and its prominent metabolite 116-N1 in Caucasian healthysubjects | Day 1,Day 5,Day 6:until 48 hours post-dose.
  Pharmacokinetic (PK) parameters: elimination half-life (t1/2) of JT001 (VV116) and its metabolite 116-N1.
To explore the pharmacokinetics of JT001 and its prominent metabolite 116-N1 in Caucasian healthysubjects | Day 1,Day 5,Day 6:until 48 hours post-dose.
  Pharmacokinetic (PK) parameters: apparent clearance (CL/F) of JT001 (VV116) and its metabolite 116-N1.
To explore the pharmacokinetics of JT001 and its prominent metabolite 116-N1 in Caucasian healthysubjects | Day 1,Day 5,Day 6:until 48 hours post-dose.
  Pharmacokinetic (PK) parameters: mean residence time (MRT) of JT001 (VV116) and its metabolite 116-N1.
To explore the pharmacokinetics of JT001 and its prominent metabolite 116-N1 in Caucasian healthysubjects | Day 1,Day 5,Day 6:until 48 hours post-dose.
  Pharmacokinetic (PK) parameters : apparent volume of distribution (Vz/F) Of JT001 (VV116) and its metabolite 116-N1.
To explore the pharmacokinetics of JT001 and its prominent metabolite 116-N1 in Caucasian healthysubjects | Day 1,Day 5,Day 6:until 48 hours post-dose.
  Pharmacokinetic (PK) parameters: accumulation ratio (Rac) of JT001 (VV116) and its metabolite 116-N1.

SECONDARY OUTCOMES:
To evaluate the safety and tolerability of JT001 tablets in Caucasian healthy subjects after multiple dosesoral administrations. | Up to 12 days
  Safety data: adverse events (AEs). AEs will be coded using the most current version of the MedDRA® Version 25.0 or higher. The numbers of cases and incidences of all TEAEs, drug-related TEAEs, SAEs, and TEAEs leading to withdrawal should be classified and summarised according to the dose group, SOC, and PT. TEAEs will also be summarised by severity and by relationship to study drug.
To evaluate the safety and tolerability of JT001 tablets in Caucasian healthy subjects after multiple dosesoral administrations. | Up to 12 days
  Safety data: vital signs, Respiration(beats per minute) The number and percentages of subjects with abnormal vital signs (respiration, blood pressure, body temperature, and pulse) will be listed and summarised by treatment and protocol specified collection time point. Observed and change from baseline will be summarised at each protocol specified collection time point by dosing group.
To evaluate the safety and tolerability of JT001 tablets in Caucasian healthy subjects after multiple dosesoral administrations. | Up to 12 days
  Safety data:vital signs,blood pressure(mm Hg) The number and percentages of subjects with abnormal vital signs (respiration, blood pressure, body temperature, and pulse) will be listed and summarised by treatment and protocol specified collection time point. Observed and change from baseline will be summarised at each protocol specified collection time point by dosing group.
To evaluate the safety and tolerability of JT001 tablets in Caucasian healthy subjects after multiple dosesoral administrations. | Up to 12 days
  Safety data:vital signs,body temperature(℃) The number and percentages of subjects with abnormal vital signs (respiration, blood pressure, body temperature, and pulse) will be listed and summarised by treatment and protocol specified collection time point. Observed and change from baseline will be summarised at each protocol specified collection time point by dosing group.
To evaluate the safety and tolerability of JT001 tablets in Caucasian healthy subjects after multiple dosesoral administrations. | Up to 12 days
  Safety data:vital signs,pulse(beats per minute) The number and percentages of subjects with abnormal vital signs (respiration, blood pressure, body temperature, and pulse) will be listed and summarised by treatment and protocol specified collection time point. Observed and change from baseline will be summarised at each protocol specified collection time point by dosing group.
To evaluate the safety and tolerability of JT001 tablets in Caucasian healthy subjects after multiple dosesoral administrations. | Up to 12 days
  Safety data: laboratory tests,The number and percentages of subjects with abnormal laboratory tests (including haematology, biochemistry, coagulation, and urinalysis) in each dose group will be summarised. All abnormal laboratory test indicators and abnormal clinically significant indicators will be listed.
To evaluate the safety and tolerability of JT001 tablets in Caucasian healthy subjects after multiple dosesoral administrations. | Up to 12 days
  Safety data: physical examinations, include general appearance, head, ears, eyes, nose, throat, dentition, thyroid, chest (heart, lungs), abdomen, skin, neurological, extremities, back, neck, musculoskeletal, and lymph nodes.
  The number and percentages of subjects with abnormal physical examination in each dose group will be summarised.
To evaluate the safety and tolerability of JT001 tablets in Caucasian healthy subjects after multiple dosesoral administrations. | Up to 12 days
  Safety data: 12-lead electrocardiograms (ECGs): heart rate. The number and percentages of subjects with abnormal ECG values will be listed and summarised by treatment by protocol specified collection time point by dosing group.
To evaluate the safety and tolerability of JT001 tablets in Caucasian healthy subjects after multiple dosesoral administrations. | Up to 12 days
  Safety data: 12-lead electrocardiograms (ECGs): P-R interval. The number and percentages of subjects with abnormal ECG values will be listed and summarised by treatment by protocol specified collection time point by dosing group.
To evaluate the safety and tolerability of JT001 tablets in Caucasian healthy subjects after multiple dosesoral administrations. | Up to 12 days
  Safety data: 12-lead electrocardiograms (ECGs): QTcF interval. The number and percentages of subjects with abnormal ECG values will be listed and summarised by treatment by protocol specified collection time point by dosing group.

CONTACTS AND LOCATIONS:
Overall Officials: Juan Ma, Master, Study Director — Shanghai Junshi Bioscience Co., Ltd.

IPD SHARING:
Plan to Share IPD: Undecided